CLINICAL TRIAL: NCT07088926
Title: A Phase IIb Randomized, Double-blind, Placebo-controlled, Parallel, Multidose Study to Evaluate the Efficacy, Safety, and PK of AZD0292 in Participants 12 Years of Age and Older With Bronchiectasis and Chronic Pseudomonas Aeruginosa Colonization
Brief Title: A Study to Evaluate the Efficacy, Safety, and PK of AZD0292 Administered IV in Participants 12 Years of Age and Older With Bronchiectasis and Chronic Pseudomonas Aeruginosa Colonization
Acronym: CLEAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D7700C00003
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Bronchiectasis With Pseudomonas Aeruginosa Colonization
Keywords: Bronchiectasis Chronic Pseudomonas Aeruginosa Colonization

STUDY DESIGN:
Intervention Model Description: D7700C00003 is a multicenter, randomized, Phase IIb, double-blind, placebo-controlled, parallel, multidose study to evaluate the efficacy, safety, and PK of AZD0292 compared with placebo in participants with bronchiectasis and chronic PsA colonization. The study will enroll up to 435 bronchiectasis participants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, Investigators, site staff, and AstraZeneca study staff who are involved in the treatment or clinical evaluation and monitoring of the participants will remain blinded to each participant's treatment assignment throughout the course of the study. As AZD0292 and placebo are visually distinct prior to dose preparation, an unblinded pharmacist (or designee, in accordance with local and institutional regulations) will be responsible for the handling and dose preparation of all study intervention and will endeavor to ensure that there are no differences in time taken to dispense following randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose (Experimental): High-Dose AZD0292 administered starting on Day 1, subsequent administrations per schedule of assessments.
  Interventions: Biological: AZD0292
- Low-dose (Experimental): Low-dose AZD0292 administered starting on Day 1, subsequent administrations per schedule of assessments.
  Interventions: Biological: AZD0292
- Placebo (Placebo Comparator): Placebo administered starting on Day 1, subsequent administrations per schedule of assessments.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AZD0292 — AZD0292 high-dose or low-dose administered starting on Day 1 via IV infusion, subsequent administrations per schedule of assessments.
  Arms: High-dose; Low-dose
Other: Placebo — Placebo administered starting on Day 1 via IV infusion, subsequent administrations per schedule of assessments.
  Arms: Placebo

SUMMARY:
AZD0292 is a bispecific IgG1k mAb being evaluated for the prevention of exacerbations in bronchiectasis patients chronically colonized with PsA.

DETAILED DESCRIPTION:
AZD0292 is a bispecific IgG1k mAb being evaluated for the prevention of exacerbations in bronchiectasis patients chronically colonized with PsA.

This Phase IIb study aims to assess the efficacy, safety, and PK of 2 dosage regimens of AZD0292 administered IV, as compared to placebo in participants 12 years of age and older.

The primary population of this study will be PsA-colonized NCFBE patients, a bronchiectasis group with frequent pulmonary exacerbations due to chronic PsA airway colonization. These PsA associated pulmonary exacerbations contribute to a decline in lung function, impair quality of life and increase mortality, highlighting the urgent need for effective therapeutic options. To investigate the broader applicability of AZD0292, bronchiectasis patients with CF who are colonized with PsA will be also included as a non-powered exploratory group in this Phase IIb study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 12 years of age at the time of signing the informed consent/assent
2. Weight ≥ 35 kg
3. Bronchiectasis diagnosed by a physician and confirmed by CT demonstrating abnormal bronchial dilation in ≥ 1 lobe. Note: A historical CT scan within the past 5 years is acceptable. If not available, a CT scan should be conducted at screening to confirm eligibility.
4. Participants who are receiving appropriate standard of care therapy per local guidelines and have a documented history of ≥ 2 moderate exacerbations or ≥ 1 severe exacerbation in the preceding 12 months requiring antibiotics
5. Participants who are clinically stable and free from an exacerbation of bronchiectasis for 4 weeks prior to randomization
6. Participants with pre- or post-bronchodilator FEV1 ≥ 25% predicted value at screening.
7. Presence of positive (PCR or culture) PsA in an airway sample at least once in the last 24 months prior to screening
8. Presence of culture positive PsA in sputum at least within 5 weeks of randomization. Participants who have previously received PsA eradication therapy, as determined appropriate by their treating provider, but remain colonized with PsA are eligible for the study.
9. Capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

1. Primary lung diagnosis other than bronchiectasis
2. Evidence of active tuberculosis or active nontuberculous mycobacteria being treated or requiring treatment. Participants currently receiving treatment for active TB or nontuberculous mycobacteria may be considered after completion of an appropriate course of therapy
3. Evidence of an active allergic bronchopulmonary aspergillosis being treated or requiring treatment
4. Need for long term supplemental oxygen. Oxygen use for ambulation and relief of breathlessness after exercise is allowed
5. Malignancy, current or within the previous 5 years, except for stable prostate cancer, adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma in situ treated with apparent success more than one year prior to enrolment
6. AIDS or Advanced human immunodeficiency virus disease (CD4 count of < 200 cells/mm3)
7. History of severe adverse reaction associated with a mAb, and/or history of severe allergic reaction (eg, anaphylaxis that required the use of epinephrine/adrenaline or hospitalization), and/or history of immune complex disease (Type III hypersensitivity reactions) to monoclonal antibody administration
8. Treatment with long term anti-PsA antibiotics, macrolides, or DPP-1 inhibitors, which are newly initiated within the 3 months prior to screening
9. Chronic immunosuppressive therapy (including prednisolone > 5 mg or equivalent) newly initiated within the last 3 months
10. Receipt of investigational products indicated for the treatment or prevention of bronchiectasis exacerbations or expected receipt during the study
11. Participants with CF on CFTR modulator therapies which are newly initiated within the previous 3 months prior to screening
12. Female participants who are pregnant, lactating, or WOCBP and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to study intervention administration and until at least 6 months after study intervention administration

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-12-09 (Estimated); Study Completion 2028-06-14 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of exacerbations over a variable follow-up time | Min 28 weeks, max 52 weeks
  To evaluate the effect of IV AZD0292 compared to placebo on the rate of moderate-to-severe pulmonary exacerbations in participants with NCFBE and chronic colonization with PsA.

SECONDARY OUTCOMES:
Annualized rate of severe exacerbations over a variable follow-up time | Min 28 weeks, max 52 weeks
  To evaluate the effect of AZD0292 compared to placebo on severe exacerbations in participants with NCFBE and chronic colonization with PsA
Change from baseline in QOL-B-RSS | Over the observation period (Week 0 to Final Dose+4 weeks)
  To evaluate the effect of AZD0292 compared to placebo on quality of life, as assessed by QoL-B-RSS over the observation period
Change from baseline in SGRQ score | Over the observation period (Week 0 to Final Dose +4 weeks)
  To evaluate the effect of AZD0292 compared to placebo on quality of life, as assessed by SGRQ over the observation period.
Time to first moderate or severe exacerbation | Through study completion (Final Dose +24 weeks)
  To evaluate the effect of AZD0292 compared to placebo on time to first pulmonary exacerbation in participants with NCFBE and chronic colonization with PsA.
Serum PK Concentrations | At specified timepoints between Week 0 and Final Dose+12 weeks
  To evaluate the PK of IV doses of AZD0292 in participants with bronchiectasis and chronic colonization with PsA
Incidence of ADA and ADA titers to AZD0292 | At specified timepoints between Week 0 and Final Dose +12 weeks
  To evaluate the immunogenicity of IV doses of AZD0292 in participants with bronchiectasis and chronic colonization with PsA
Incidence of AEs, SAEs, AESIs and MAAEs | Occurrence of AEs; first dose through 12 weeks after last study intervention administration. Occurrence of SAEs, AESIs, and MAAEs; through study completion (Final Dose+24 weeks)
  To assess the safety of AZD0292 compared with placebo in participants with bronchiectasis and chronic colonization with PsA

CONTACTS AND LOCATIONS:
Locations (142):
- United States (21):
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Plantation, Florida
  - Research Site, Rincon, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Tulsa, Oklahoma
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Mansfield, Texas
- Argentina (4):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Florida
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Australia (2):
  - Research Site, Macquarie University
  - Research Site, South Brisbane
- Belgium (4):
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Sint-Niklaas
- Brazil (7):
  - Research Site, Blumenau
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São José dos Campos
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (4):
  - Research Site, Concepción
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Viña del Mar
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
  - Research Site, Odense C
  - Research Site, Roskilde
- France (8):
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (8):
  - Research Site, Darmstadt
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Konstanz
  - Research Site, München
  - Research Site, München-Pasing
- Greece (5):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (7):
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torrette
- Research Site, Kiyose-shi, Japan
- Malaysia (3):
  - Research Site, Bandar Puncak Alam
  - Research Site, Kuala Lumpur
  - Research Site, Sibu
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
  - Research Site, Zutphens
- Peru (2):
  - Research Site, Bellavista
  - Research Site, Lima
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, Tondo
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Patraix
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bang Kra So
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Pathum Thani
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Mersin
  - Research Site, Zeytinburnu
- United Kingdom (9):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Brighton
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Liverpool
  - Research Site, Manchester
- Vietnam (6):
  - Research Site, Can Tho
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Araujo D, Shteinberg M, Aliberti S, Goeminne PC, Hill AT, Fardon TC, Obradovic D, Stone G, Trautmann M, Davis A, Dimakou K, Polverino E, De Soyza A, McDonnell MJ, Chalmers JD. The independent contribution of Pseudomonas aeruginosa infection to long-term clinical outcomes in bronchiectasis. Eur Respir J. 2018 Jan 31;51(2):1701953. doi: 10.1183/13993003.01953-2017. Print 2018 Feb. PMID 29386336
- [Background] Artaraz A, Crichton ML, Finch S, Abo-Leyah H, Goeminne P, Aliberti S, Fardon T, Chalmers JD. Development and initial validation of the bronchiectasis exacerbation and symptom tool (BEST). Respir Res. 2020 Jan 13;21(1):18. doi: 10.1186/s12931-019-1272-y. PMID 31931782
- [Background] Bellelli G, Chalmers JD, Sotgiu G, Dore S, McDonnell MJ, Goeminne PC, Dimakou K, Skrbic D, Lombi A, Pane F, Obradovic D, Fardon TC, Rutherford RM, Pesci A, Aliberti S. Characterization of bronchiectasis in the elderly. Respir Med. 2016 Oct;119:13-19. doi: 10.1016/j.rmed.2016.08.008. Epub 2016 Aug 17. PMID 27692133
- [Background] CFFPR 2023 Cystic Fibrosis Foundation Patient Registry. Bethesda, MD. 2023 Annual Data Report. Available at https://www.cff.org/media/34491/download.
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Chalmers JD, Aliberti S, Blasi F. Management of bronchiectasis in adults. Eur Respir J. 2015 May;45(5):1446-62. doi: 10.1183/09031936.00119114. Epub 2015 Mar 18. PMID 25792635
- [Background] Chalmers JD, Chang AB, Chotirmall SH, Dhar R, McShane PJ. Bronchiectasis. Nat Rev Dis Primers. 2018 Nov 15;4(1):45. doi: 10.1038/s41572-018-0042-3. PMID 30442957
- [Background] Chalmers JD, Aliberti S, Filonenko A, Shteinberg M, Goeminne PC, Hill AT, Fardon TC, Obradovic D, Gerlinger C, Sotgiu G, Operschall E, Rutherford RM, Dimakou K, Polverino E, De Soyza A, McDonnell MJ. Characterization of the "Frequent Exacerbator Phenotype" in Bronchiectasis. Am J Respir Crit Care Med. 2018 Jun 1;197(11):1410-1420. doi: 10.1164/rccm.201711-2202OC. PMID 29357265
- [Background] Chalmers JD, Chotirmall SH. Bronchiectasis: new therapies and new perspectives. Lancet Respir Med. 2018 Sep;6(9):715-726. doi: 10.1016/S2213-2600(18)30053-5. Epub 2018 Feb 23. PMID 29478908
- [Background] Chawla K, Vishwanath S, Manu MK, Lazer B. Influence of pseudomonas aeruginosa on exacerbation in patients with bronchiectasis. J Glob Infect Dis. 2015 Jan-Mar;7(1):18-22. doi: 10.4103/0974-777X.150885. PMID 25722615
- [Background] Choate R, Aksamit TR, Mannino D, Addrizzo-Harris D, Barker A, Basavaraj A, Daley CL, Daniels MLA, Eden E, DiMango A, Fennelly K, Griffith DE, Johnson MM, Knowles MR, McShane PJ, Metersky ML, Noone PG, O'Donnell AE, Olivier KN, Salathe MA, Schmid A, Thomashow B, Tino G, Winthrop KL, Stone G. Pseudomonas aeruginosa associated with severity of non-cystic fibrosis bronchiectasis measured by the modified bronchiectasis severity score (BSI) and the FACED: The US bronchiectasis and NTM Research Registry (BRR) study. Respir Med. 2021 Feb;177:106285. doi: 10.1016/j.rmed.2020.106285. Epub 2020 Dec 24. PMID 33401148
- [Background] Choi H, Xu JF, Chotirmall SH, Chalmers JD, Morgan LC, Dhar R. Bronchiectasis in Asia: a review of current status and challenges. Eur Respir Rev. 2024 Sep 25;33(173):240096. doi: 10.1183/16000617.0096-2024. Print 2024 Jul. PMID 39322263
- [Background] Ciofu O, Tolker-Nielsen T. Tolerance and Resistance of Pseudomonas aeruginosa Biofilms to Antimicrobial Agents-How P. aeruginosa Can Escape Antibiotics. Front Microbiol. 2019 May 3;10:913. doi: 10.3389/fmicb.2019.00913. eCollection 2019. PMID 31130925
- [Background] DiGiandomenico A, Warrener P, Hamilton M, Guillard S, Ravn P, Minter R, Camara MM, Venkatraman V, Macgill RS, Lin J, Wang Q, Keller AE, Bonnell JC, Tomich M, Jermutus L, McCarthy MP, Melnick DA, Suzich JA, Stover CK. Identification of broadly protective human antibodies to Pseudomonas aeruginosa exopolysaccharide Psl by phenotypic screening. J Exp Med. 2012 Jul 2;209(7):1273-87. doi: 10.1084/jem.20120033. Epub 2012 Jun 25. PMID 22734046
- [Background] Emerson J, Rosenfeld M, McNamara S, Ramsey B, Gibson RL. Pseudomonas aeruginosa and other predictors of mortality and morbidity in young children with cystic fibrosis. Pediatr Pulmonol. 2002 Aug;34(2):91-100. doi: 10.1002/ppul.10127. PMID 12112774
- [Background] FLETCHER CM, ELMES PC, FAIRBAIRN AS, WOOD CH. The significance of respiratory symptoms and the diagnosis of chronic bronchitis in a working population. Br Med J. 1959 Aug 29;2(5147):257-66. doi: 10.1136/bmj.2.5147.257. No abstract available. PMID 13823475
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Guo J, Garratt A, Hill A. Worldwide rates of diagnosis and effective treatment for cystic fibrosis. J Cyst Fibros. 2022 May;21(3):456-462. doi: 10.1016/j.jcf.2022.01.009. Epub 2022 Feb 4. PMID 35125294
- [Background] Harrington NE, Kottara A, Cagney K, Shepherd MJ, Grimsey EM, Fu T, Hull RC, Chong CE, Baker KS, Childs DZ, Fothergill JL, Chalmers JD, Brockhurst MA, Paterson S. Global genomic diversity of Pseudomonas aeruginosa in bronchiectasis. J Infect. 2024 Nov;89(5):106275. doi: 10.1016/j.jinf.2024.106275. Epub 2024 Sep 16. PMID 39293722
- [Background] Hill AT, Haworth CS, Aliberti S, Barker A, Blasi F, Boersma W, Chalmers JD, De Soyza A, Dimakou K, Elborn JS, Feldman C, Flume P, Goeminne PC, Loebinger MR, Menendez R, Morgan L, Murris M, Polverino E, Quittner A, Ringshausen FC, Tino G, Torres A, Vendrell M, Welte T, Wilson R, Wong C, O'Donnell A, Aksamit T; EMBARC/BRR definitions working group. Pulmonary exacerbation in adults with bronchiectasis: a consensus definition for clinical research. Eur Respir J. 2017 Jun 8;49(6):1700051. doi: 10.1183/13993003.00051-2017. Print 2017 Jun. PMID 28596426
- [Background] Horcajada JP, Montero M, Oliver A, Sorli L, Luque S, Gomez-Zorrilla S, Benito N, Grau S. Epidemiology and Treatment of Multidrug-Resistant and Extensively Drug-Resistant Pseudomonas aeruginosa Infections. Clin Microbiol Rev. 2019 Aug 28;32(4):e00031-19. doi: 10.1128/CMR.00031-19. Print 2019 Sep 18. PMID 31462403
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Jones 2022 Jones P. St George's Respiratory Questionnaire Manual. Version 2.4. St George's University of London. March 2022. Available at https://www.sgul.ac.uk/research/researchoperations/ research-administration/st-georges-respiratory-questionnaire/docs/SGRQ-Manual- March-2022.pdf.
- [Background] Laska IF, Crichton ML, Shoemark A, Chalmers JD. The efficacy and safety of inhaled antibiotics for the treatment of bronchiectasis in adults: a systematic review and meta-analysis. Lancet Respir Med. 2019 Oct;7(10):855-869. doi: 10.1016/S2213-2600(19)30185-7. Epub 2019 Aug 9. PMID 31405826
- [Background] Long MB, Gilmour A, Kehl M, Tabor DE, Keller AE, Warrener P, Gopalakrishnan V, Rosengren S, Crichton ML, McIntosh E, Giam YH, Keir HR, Brailsford W, Hughes R, Belvisi MG, Sellman BR, DiGiandomenico A, Chalmers JD. A Bispecific Monoclonal Antibody Targeting Psl and PcrV Enhances Neutrophil-Mediated Killing of Pseudomonas aeruginosa in Patients with Bronchiectasis. Am J Respir Crit Care Med. 2024 Jul 1;210(1):35-46. doi: 10.1164/rccm.202308-1403OC. PMID 38754132
- [Background] Long et al 2025 Long MB, Hull RC, Gilmour A, Viligorska K, Richardson H, New BJM, et al. A bispecific monoclonal antibody targeting Psl and PcrV for chronic pseudomonas aeruginosa infection in patients With bronchiectasis: results From a randomized, double-blind placebo-controlled trial (GREAT-2) [abstract]. Am J Respir Crit Care Med 2025;211:A3117.
- [Background] Nigro M, Laska IF, Traversi L, Simonetta E, Polverino E. Epidemiology of bronchiectasis. Eur Respir Rev. 2024 Oct 9;33(174):240091. doi: 10.1183/16000617.0091-2024. Print 2024 Oct. PMID 39384303
- [Background] O'Donnell AE. Bronchiectasis - A Clinical Review. N Engl J Med. 2022 Aug 11;387(6):533-545. doi: 10.1056/NEJMra2202819. No abstract available. PMID 35947710
- [Background] Oswalt ML, Kemp SF. Anaphylaxis: office management and prevention. Immunol Allergy Clin North Am. 2007 May;27(2):177-91, vi. doi: 10.1016/j.iac.2007.03.004. PMID 17493497
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Quittner AL, Marciel KK, Salathe MA, O'Donnell AE, Gotfried MH, Ilowite JS, Metersky ML, Flume PA, Lewis SA, McKevitt M, Montgomery AB, O'Riordan TG, Barker AF. A preliminary quality of life questionnaire-bronchiectasis: a patient-reported outcome measure for bronchiectasis. Chest. 2014 Aug;146(2):437-448. doi: 10.1378/chest.13-1891. PMID 24626872
- [Background] Quittner AL, O'Donnell AE, Salathe MA, Lewis SA, Li X, Montgomery AB, O'Riordan TG, Barker AF. Quality of Life Questionnaire-Bronchiectasis: final psychometric analyses and determination of minimal important difference scores. Thorax. 2015 Jan;70(1):12-20. doi: 10.1136/thoraxjnl-2014-205918. Epub 2014 Oct 16. PMID 25323621
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Background] Sibila O, Laserna E, Shoemark A, Keir HR, Finch S, Rodrigo-Troyano A, Perea L, Lonergan M, Goeminne PC, Chalmers JD. Airway Bacterial Load and Inhaled Antibiotic Response in Bronchiectasis. Am J Respir Crit Care Med. 2019 Jul 1;200(1):33-41. doi: 10.1164/rccm.201809-1651OC. PMID 31109172
- [Background] Song J, Sin S, Kang HR, Oh YM, Jeong I; KMBARC. Clinical Impacts of Pseudomonas aeruginosa Isolation in Patients with Bronchiectasis: Findings from KMBARC Registry. J Clin Med. 2024 Aug 24;13(17):5011. doi: 10.3390/jcm13175011. PMID 39274224
- [Background] Tabor DE, Oganesyan V, Keller AE, Yu L, McLaughlin RE, Song E, Warrener P, Rosenthal K, Esser M, Qi Y, Ruzin A, Stover CK, DiGiandomenico A. Pseudomonas aeruginosa PcrV and Psl, the Molecular Targets of Bispecific Antibody MEDI3902, Are Conserved Among Diverse Global Clinical Isolates. J Infect Dis. 2018 Nov 5;218(12):1983-1994. doi: 10.1093/infdis/jiy438. PMID 30016475
- [Background] Tomaszewski EL, Atkinson MJ, Janson C, Karlsson N, Make B, Price D, Reddel HK, Vogelmeier CF, Mullerova H, Jones PW; NOVELTY Scientific Community; NOVELTY study investigators. Chronic Airways Assessment Test: psychometric properties in patients with asthma and/or COPD. Respir Res. 2023 Apr 8;24(1):106. doi: 10.1186/s12931-023-02394-6. PMID 37031164
- [Background] WHO 2017 WHO. WHO/EMP/IAU/2017.12 Prioritization of pathogens to guide discovery, research and development of new antibiotics for drug-resistant bacterial infections, including tuberculosis. Report. World Health Organization, WHO, Antimicrobial Resistance Division Global Coordination and Partnership, Medicines Selection, IP and Affordability. Available from: http://www.who.int/publications/i/item/WHO-EMP-IAU-2017.02.
- [Background] Wilson R, Aksamit T, Aliberti S, De Soyza A, Elborn JS, Goeminne P, Hill AT, Menendez R, Polverino E. Challenges in managing Pseudomonas aeruginosa in non-cystic fibrosis bronchiectasis. Respir Med. 2016 Aug;117:179-89. doi: 10.1016/j.rmed.2016.06.007. Epub 2016 Jun 7. PMID 27492530
- [Background] Zolin et al 2024 Zolin A, Adamoli A, Bakkeheim E, van Rens J, et al. ECFSPR Annual Report 2022. Published 2024. Available at https://www.ecfs.eu/sites/default/files/Annual%20Report_2022_ECFSPR_20240603.pdf.